CLINICAL TRIAL: NCT06045364
Title: Effect of Glycopyrrolate on Nausea and Vomiting After ERCP Operation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jie Chen (Other)
Responsible Party: Sponsor-Investigator, Jie Chen, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-115
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Glycopyrrolate; anisodamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycopyrrolate (Experimental): During induction of anesthesia, 0.2mg Glycopyrrolate was given intravenously to participants.
  Interventions: Drug: Glycopyrrolate
- Anisodamine Group (Active Comparator): During induction of anesthesia,10mg of Anisodamine was given intramuscular injection
  Interventions: Drug: Anisodamine

INTERVENTIONS:
Drug: Glycopyrrolate — During induction of anesthesia, 0.2mg Glycopyrrolate was given intravenously
  Arms: Glycopyrrolate
Drug: Anisodamine — During induction of anesthesia,10mg of Anisodamine was given intramuscular injection.
  Arms: Anisodamine Group

SUMMARY:
This study aims to determine the role of Glycopyrrolate in preventing postoperative nausea and vomiting of ERCP.

DETAILED DESCRIPTION:
This study is a prospective, double-blind, randomized controlled trial. Patients who meet the criteria of our center and need to undergo ERCP lesion resection will be included and randomly divided into groups. After receiving Glycopyrrolate (experimental group) and Anisodamine (control group), duodenal peristalsis, biliary and pancreatic treatment time and postoperative nausea and vomiting will be observed during therapeutic ERCP. The inhibitory effect of Glycopyrrolate on postoperative nausea and vomiting of ERCP will be analyzed statistically.

Main outcome measure: incidence of nausea and vomiting after ERCP Secondary outcome measures: mean duodenal contractions per minute, duodenal spasm frequency and score, ERCP operation time, occurrence of other side effects of medication, remedial medication, and incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* 1.Adults 18-80 years old 2.ASA :I-III 3.Patients who are able to give informed consent and are currently planning to have the lesion removed or examined at the descending ERCP

Exclusion Criteria:1: Use of anticholinergic drugs

2: pregnancy

3: glaucoma

4: Myasthenia gravis

5: Obstructive gastrointestinal diseases

6: Obstructive urinary tract disease (prostatic hyperplasia)

7: Heart disease (coronary heart disease, congestive heart failure)

8: hyperthyroidism

9: Previous history of abdominal or intestinal surgery

10: Chronic renal failure

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | Timepoint：24 hours after the ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, doctor, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No